CLINICAL TRIAL: NCT02213679
Title: Guanidinoacetic Acid Loading for Chronic Fatigue Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Health Sciences, Serbia (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Sergej M. Ostojic, MD, PhD, Associate Professor of Biomedical Sciences, Center for Health Sciences, Serbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 878/13-EUTC:03
Record Dates: First submitted 2014-08-05; First posted 2014-08-11 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Fatigue Syndrome
Keywords: Creatine; Guanidinoacetic acid; Intervention; Fatigue; Muscle strength
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue | interventions — glycocyamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guanidinoacetic acid (Experimental): Supplementation with dietary guanidinoacetic acid
  Interventions: Dietary Supplement: Guanidinoacetic acid
- Placebo (Placebo Comparator): Supplementation with cellulose
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Guanidinoacetic acid — Dietary supplement
  Arms: Guanidinoacetic acid
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Chronic fatigue syndrome (CFS) is a debilitating condition of unknown etiology. Recent studies have shown that CFS is associated with impaired cellular energetics and low levels of phosphocreatine. Since guanidinoacetic acid (GAA) acts as a highly bioavailable precursor of creatine it may provide an ideal dietary supplement to facilitate treatment and perhaps prevention of CFS. The overall hypothesis to be evaluated is that medium-term supplementation with GAA will improve clinical outcomes in well-defined adult CFS patients via augmented provision of creatine. Specific aims: (1) To determine the effects of GAA on CFS symptomatology using a fatigue severity inventory, soreness of locomotive apparatus scales, and a health-related quality of life survey; (2) To determine the effect of GAA on creatine metabolism using laboratory studies and magnetic resonance spectroscopy; (3) To characterize the physiological effects of GAA on work capacity via actigraphy and exercise performance tests; and (4); To determine the prevalence of subjectively reported side-effects and biochemical adverse events associated with GAA intervention.

DETAILED DESCRIPTION:
A variety of dietary interventions have been used in the management of CFS, yet no therapeutic modality demonstrated overall positive results in terms of effectiveness (Whiting et al. 2001). Previous studies have evaluated the effects of essential fatty acids, vitamins, minerals and/or enzymes, with findings do not support the use of a broad-spectrum nutritional supplement in treating CFS-related symptoms (Brouwers et al. 2002). Considering the fact that patients with CFS have lower levels of high-energy compounds (e.g. phosphocreatine, adenosine triphosphate) (Block et al. 1998), effective dietary treatment of CFS should be focused on providing compounds that facilitates cellular bioenergetics. Besides other candidate agents, guanidinoacetic acid (GAA) could be of particular interest since it occurs naturally in the human body and acts as an immediate precursor of creatine (Wyss and Kaddurah-Daouk, 2000). Due to its low cost and high bioavailability (Baker 2009), if proven effective dietary GAA may be suitable for use in broad CFS population.

ELIGIBILITY:
Inclusion Criteria:

* Adults who fulfilled the 1994 CDC criteria for CFS
* Older than 18 years of age will be candidates for inclusion in the study.

Exclusion Criteria:

* Psychiatric comorbidity
* Use of any dietary supplement within 4-weeks prior to the study commencing
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in the Multidimensional Fatigue Inventory (MFI) score | Baseline and afetr 3 months

SECONDARY OUTCOMES:
Pain in the locomotive apparatus | Baseline and after 3 months

OTHER OUTCOMES:
Health-related quality of life | Baseline and after 3 months
Daily physical activity | Baseline and after 3 months
  Measurement of duration, frequency, and intensity of various types of human physical activity (exercise and nonexercise physical activity)
Muscular strength | Baseline and after 3 months
  For muscular performance, maximal voluntary strength of knee extensor muscles will be measured bilaterally using an isometric dynamometer during static knee joint movement with leg at 165º of flexion (180º = leg fully extended). The better of two efforts for each leg will be recorded with cumulative value presented as total isometric strength.
Serum creatine | Baseline and after 3 months
Side-effects prevalence | During 3 months of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sergej M Ostojic, MD, PhD, Principal Investigator — Faculty of Sport and Physical Education, Novi Sad
Locations (1):
- Center for Health, Exercise and Sport Sciences, Belgrade, Serbia, Serbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ostojic SM, Niess B, Stojanovic M, Obrenovic M. Creatine metabolism and safety profiles after six-week oral guanidinoacetic acid administration in healthy humans. Int J Med Sci. 2013;10(2):141-7. doi: 10.7150/ijms.5125. Epub 2013 Jan 3. PMID 23329885
- [Background] Ostojic SM, Niess B, Stojanovic M, Obrenovic M. Co-administration of methyl donors along with guanidinoacetic acid reduces the incidence of hyperhomocysteinaemia compared with guanidinoacetic acid administration alone. Br J Nutr. 2013 Sep 14;110(5):865-70. doi: 10.1017/S0007114512005879. Epub 2013 Jan 28. PMID 23351309
- [Background] Ostojic SM, Stojanovic M, Drid P, Hoffman JR. Dose-response effects of oral guanidinoacetic acid on serum creatine, homocysteine and B vitamins levels. Eur J Nutr. 2014 Dec;53(8):1637-43. doi: 10.1007/s00394-014-0669-0. Epub 2014 Feb 18. PMID 24535415